CLINICAL TRIAL: NCT06041529
Title: An Open-Label, Superiority, Randomized, Comparative Study to Evaluate the Efficacy and Safety of Telmisartan, Amlodipine, and Chlorthalidone Fixed-Dose Combination Versus Telmisartan, Amlodipine, and Hydrochlorothiazide in Elderly Patients with Essential Hypertension Uncontrolled by Telmisartan and Amlodipine Combinations
Brief Title: Study to Evaluate the Efficacy and Safety of TEL/AML/CTD in Elderly Patients with Essential Hypertension
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC050
Record Dates: First submitted 2023-09-04; First posted 2023-09-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Essential Hypertension
Keywords: Telmisartan/Amlodipine/Chlorthalidone Fixed-Dose Combination
MeSH Terms: conditions — Essential Hypertension | interventions — Telmisartan; Amlodipine; Chlorthalidone; Hydrochlorothiazide; telmisartan amlodipine combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telmisartan/Amlodipine/Chlorthalidonea 40/5/12.5 mg (Experimental): Telmisartan/Amlodipine/Chlorthalidonea 40/5/12.5 mg will be orally administered during the study period
  Interventions: Drug: Telmisartan/Amlodipine/Chlorthalidone 40/5/12.5 mg
- Telmisartan/Amlodipine/Hydrochlorothiazide 40/5/25 mg (Active Comparator): Telmisartan/Amlodipine 40/5 mg and Hydrochlorothiazide 25 mg will be orally administered each during study period
  Interventions: Drug: Telmisartan/Amlodipine/Hydrochlorothiazide 40/5/25 mg

INTERVENTIONS:
Drug: Telmisartan/Amlodipine/Chlorthalidone 40/5/12.5 mg — PO, Once daily(QD), 8 weeks and 26 weeks if applicable
  Other Names: Truset 40/5/12.5mg
  Arms: Telmisartan/Amlodipine/Chlorthalidonea 40/5/12.5 mg
Drug: Telmisartan/Amlodipine/Hydrochlorothiazide 40/5/25 mg — PO, Once daily(QD), 8 weeks and 26 weeks if applicable
  Other Names: Twynsta 40/5 mg, Dichlozid 25 mg
  Arms: Telmisartan/Amlodipine/Hydrochlorothiazide 40/5/25 mg

SUMMARY:
This study is to compare the efficacy and safety of Telmisartan, Amlodipine, and Chlorthalidone Fixed-Dose Combination and Telmisartan, Amlodipine, and Hydrochlorothiazide in Elderly Patients with Essential Hypertension Uncontrolled by Telmisartan and Amlodipine Combinations

DETAILED DESCRIPTION:
This is a Phase IV, Randomized, Open-label, Superiority, Comparative study evaluating the efficacy and safety of Telmisartan, Amlodipine, and Chlorthalidone Fixed-Dose Combination) versus Telmisartan, Amlodipine, and Hydrochlorothiazide in eledrly patient with essential hypertension uncontrolled by Telmisartan and Amlodipine Combinations.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have been fully informed about the purpose, content, and characteristics of investigational product, and have voluntarily agreed in writing
2. Aged ≥ 65 with essential hypertension
3. Patient with uncontrolled essential hypertension at screening

   * If already taking antihypertensive drugs, mean sitting systolic blood pressure (MSSBP) must be 140 mmHg ≤ MSSBP < 200 mmHg
   * If not taking any antihypertensive drugs at least 4 weeks, mean sitting systolic blood pressure (MSSBP) must be 160 mmHg ≤ MSSBP < 200 mmHg

Exclusion Criteria:

1. Patient who has history of drug allergic reactions
2. Known hypersensitivity to components of the investigational product
3. Patient who is unable to stop taking prohibited drugs
4. Test results showing the following values at screening

   * The change of MSSBP ≥ 20 mmHg and MSDBP ≥ 10 mmHg on target arm between 1st and 2nd measurements
5. Pregnant or lactating women
6. Patient who is unable to maintain proper night sleep
7. Malnutrition, starvation, debilitating factors, A person who is being forcibly detained for the treatment of mental or physical
8. Administration of other investigational products within 3 months prior to screening.
9. An impossible one who participates in clinical trial by investigator's decision

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-06-24 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Mean Systolic Blood Pressure (MSBP) in nighttime | Week 8
  To evaluate change from baseline in nighttime Mean Systolic Blood Pressure (MSBP) measured by Ambulatory Blood Pressure Monitoring at Week 8

SECONDARY OUTCOMES:
Mean Systolic Blood Pressure (MSBP) in nighttime | Week 26 if applicable
  To evaluate change from baseline in nighttime Mean Systolic Blood Pressure (MSBP) measured by Ambulatory Blood Pressure Monitoring at Week 26 if applicable
Mean Diastolic Blood Pressure (MDBP) in nighttime | Week 8 and Week 26 if applicable
  To evaluate change from baseline in nighttime Mean Diastolic Blood Pressure (MDBP) measured by Ambulatory Blood Pressure Monitoring at Week 8 and Week 26 if applicable
Mean Systolic Blood Pressure (MSBP)/Mean Diastolic Blood Pressure (MDBP) in daytime | Week 8 and Week 26 if applicable
  To evaluate change from baseline in daytime Mean Systolic Blood Pressure (MSBP)/Mean Diastolic Blood Pressure (MDBP) measured by Ambulatory Blood Pressure Monitoring at Week 8 and Week 26 if applicable
24-hour Mean Systolic Blood Pressure (MSBP)/Mean Diastolic Blood Pressure (MDBP) | Week 8 and Week 26 if applicable
  To evaluate change from baseline in 24-hour Mean Systolic Blood Pressure (MSBP)/Mean Diastolic Blood Pressure (MDBP) measured by Ambulatory Blood Pressure Monitoring at Week 8 and Week 26 if applicable
Patients Achieving in nighttime Mean Systolic Blood Pressure (MSBP) | Week 8
  To evaluate the percentage of patients who reached the treatment goal for nighttime Mean Systolic Blood Pressure (MSBP) (<110/65mmHg) measured by Ambulatory Blood Pressure Monitoring at Week 8
Mean Sitting Systolic Blood Pressure (MSSBP)/ Mean Sitting Diastolic Blood Pressure (MSDBP) | Week 4, Week 8 and Week 26 if applicable
  To evaluate change from baseline in Mean Sitting Systolic Blood Pressure (MSSBP)/ Mean Sitting Diastolic Blood Pressure (MSDBP) measured by the Institution at Week 4, Week 8 and Week 26 if applicable
Patients Achieving in Mean Sitting Systolic Blood Pressure (MSSBP) | Week 4, Week 8 and Week 26 if applicable
  - To evaluate the percentage of patients who reached the treatment goal for Mean Sitting Blood Pressure (MSBP) < 140/90 mmHg measured by the Institution at Week 4, Week 8 and Week 26 if applicable
Percentage of patients with decreased Mean Sitting Systolic Blood Pressure (MSSBP) and Mean Sitting Diastolic Blood Pressure (MSDBP). | Week 4, Week 8 and Week 26 if applicable
  To evaluate the percentage of subjects with a Mean Sitting Systolic Blood Pressure (MSSBP) decrease of ≥20mmHg and a Mean Sitting Diastolic Blood Pressure (MSDBP) decrease of ≥10mmHg at Week 4, Week 8 and Week 26 if applicable
T/P ratio | Week 8 and Week 26 if applicable
  To evaluate the T/P ratio for systolic/diastolic blood pressure measured by Ambulatory Blood Pressure Monitoring at Week 8 and Week 26 if applicable

CONTACTS AND LOCATIONS:
Overall Officials: Sanghyun Ihm, Principal Investigator — The Catholic University of Korea Bucheon St.Mary's Hospital
Locations (15):
- South Korea (15):
  - The Catholic University of Korea Bucheon St.Mary's Hospital, Seoul, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Busan
  - The Catholic University of Korea Daejeon ST. Mary's Hospital, Daejeon
  - Wonju Severance Christian Hospital, Gangwon-do
  - Chonnam National University Hospital, Gwangju
  - Gwangju Veterans Hospital, Gwangju
  - The Catholic University of Korea, ST. Vincent's Hospital, Gyeonggi-do
  - he Catholic University of Korea, Incheon ST. Mary's Hospital, Incheon
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Hanyang university medical center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido ST. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital, Seoul
  - Seoul national University Budang hospital, Seoul

IPD SHARING:
Plan to Share IPD: No